CLINICAL TRIAL: NCT00787813
Title: Effect of Oral N-Acetyl Cysteine on Pregnancy Outcome After Cervical Cerclage: a Randomized Controlled Trial
Brief Title: N-Acetyl Cysteine After Cervical Cerclage
Acronym: NAC-CC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Prof. Ezat Hamed Sayed, Department of Obstetrics & Gynecology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NAC after cerclage
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Last update posted 2008-11-20 (Estimated); Status verified 2008-11

CONDITIONS: Cervical Cerclage
Keywords: N-acetyl cysteine (NAC); Cervical cerclage; cervical cerclage for cervical insufficiency
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): N-Acetyl Cysteine
  Interventions: Drug: N-Acetyl Cysteine
- 2 (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-Acetyl Cysteine — oral daily dose of 0.6 g of N-acetyl cysteine in effervescent form
  Other Names: placebo
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The aim of the study is to evaluate the effect of N-acetyl cysteine (NAC) on pregnancy outcome in women undergoing cervical cerclage for cervical insufficiency.

DETAILED DESCRIPTION:
A randomized controlled clinical trial to be carried out in a university-affiliated tertiary center.Participating women will be randomized into two groups: Group A will be given an oral daily dose of 0.6 g of NAC in effervescent form; group B, serving as controls, will not receive NAC.The two groups will then be compared according to pregnancy outcome.

ELIGIBILITY:
Inclusion Criteria:

* women with history suggestive of cervical insufficiency together with ultrasound findings suggestive of cervical insufficiency undergoing elective cervical cerclage between the 11th and 12th gestational week.
* singelton viable fetus

Exclusion Criteria:

* women tested positive for bacterial vaginosis
* women currently with threatened abortion (vaginal bleeding or uterinecramps)
* age older than 35 years or younger than 20 years
* unwillingness to participate
* irregular and/or uncertain menstrual dates
* rupture of membranes
* previous cesarean delivery
* possible risks for preterm birth in the current or previous pregnancy such as twin pregnancy, IUFD, malpresentation, known fetal anomaly, progesterone or heparin treatment during the current pregnancy, hypertension, and/or seizure disorders.
* women with contra indications for cervical cerclage or anesthesia.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Gestational age at delivery | 3-6 months

SECONDARY OUTCOMES:
Take home babies, neonatal morbidity | 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: AHMED M NASR, MD, Principal Investigator — Women's Health Center, Assiut University, EGYPT
Locations (1):
- Women's Health Center, Asyut, Asyut Governorate, Egypt

REFERENCES:
- [Background] Shahin AY, Hassanin IM, Ismail AM, Kruessel JS, Hirchenhain J. Effect of oral N-acetyl cysteine on recurrent preterm labor following treatment for bacterial vaginosis. Int J Gynaecol Obstet. 2009 Jan;104(1):44-8. doi: 10.1016/j.ijgo.2008.08.026. Epub 2008 Oct 11. PMID 18851855
- [Derived] Eleje GU, Eke AC, Ikechebelu JI, Ezebialu IU, Okam PC, Ilika CP. Cervical stitch (cerclage) in combination with other treatments for preventing spontaneous preterm birth in singleton pregnancies. Cochrane Database Syst Rev. 2020 Sep 24;9(9):CD012871. doi: 10.1002/14651858.CD012871.pub2. PMID 32970845